CLINICAL TRIAL: NCT00300586
Title: A Randomized Phase III Trial Assessing in Patients With Advanced Non-small Cell Lung Cancer Not Progressing on First Line Cisplatin-gemcitabine Chemotherapy Maintenance Chemotherapy With Gemcitabine or Sequential Treatment With Erlotinib
Brief Title: IFCT-GFPC 05.02 A Randomized Phase III Trial Assessing in Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005.386
Record Dates: First submitted 2006-03-06; First posted 2006-03-09 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2011-12

CONDITIONS: Stage IV Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer ;; metastatic ;; chemotherapy ;; erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Observation; Gemcitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (supervision) (Sham Comparator): medical supervision, second line chemotherapy if progression
  Interventions: Drug: observation
- B (gemcitabicine) (Active Comparator): Maintenance treatment (gemcitabicine 1250 mg/m² J1, J8 (repeated cycles every 21 days), second line chemotherapy if progression
  Interventions: Drug: gemcitabine
- C (Erlotinib) (Experimental): Treatment by erlotinib 150 mg/day (sequential treatment), second line chemotherapy if progression
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: observation — observation, second line chemotherapy if progression
  Arms: A (supervision)
Drug: gemcitabine — 1250 mg/m² D1, D8 q21 days
  Arms: B (gemcitabicine)
Drug: erlotinib — 150 mg daily
  Arms: C (Erlotinib)

SUMMARY:
The objective of this trial is to improve the duration of control disease for PS 0-1 patients who are not progressing on first-line cisplatin-gemcitabine chemotherapy. Standard therapy is for these patients to stop first-line chemotherapy after 4 to 6 cycles and to begin a second-line chemotherapy when progression of disease is occurring. Two approaches will be experimented in this trial in attempt to prolong progression free survival :

* Maintenance chemotherapy with single-agent gemcitabine continued till disease progression or toxicity.
* Sequential treatment with erlotinib immediately given after the end of first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented NSCLC (tumor tissue samples will be provided to look for assessment of EGFR status with CISH, immunochemistry and mutations) : adenocarcinoma, squamous cell carcinoma, large cell carcinoma. A cytological documentation of NSCLC is accepted.
* Stage IV disease or metastatic relapse in not previously irradiated areas of a NSCLC previously treated with surgery or radiation therapy (with a histologically documented proof of relapse) or stage III B with documented pleural involvement.
* Measurable disease according to the RECIST criteria.
* Prior radiotherapy authorized except for irradiation concerning measurable disease.
* Age >18 and < 70 years.
* PS < 2.
* Normal hepatic function : serum bilirubin < 1.5 ULN, SGOT (ASAT) and SGPT (ALAT) < 2,5 ULN ; in presence of liver metastases, SGOT and SGPT must be < 5 x ULN.
* Creatinine clearance > 60 mL/min.
* Granulocyte count > 1,5 giga/L, platelet count > 100 giga/L.
* Life expectancy > 12 weeks.
* Written (signed) informed consent for use of tumors samples.
* Written (signed) informed consent to participate in the sudy.

Exclusion Criteria:

* Small cell lung cancer, bronchiolo-alveolar carcinoma, neuro-endocrine carcinoma.
* PS > 1.
* Prior chemotherapy other than cisplatin-gemcitabine.
* Prior therapy with EGFR inhibitor (e.g. monoclonal antibody).
* No concomitant therapy with phenytoin, carbamazepine, rifampicine or phenobarbital.
* Concomitant radiotherapy except for localized bone irradiation.
* Symptomatic brain metastases.
* Superior vena cava syndrome.
* Any unstable systemic disease : significant cardiovascular disease including myocardial infarction within the previous year, active infection, significant hepatic or renal disease.
* Pre-existing interstitial lung disease.
* Any inflammatory changes of the surface of the eyes.
* Psychiatric disease with inability to understand the study or to comply with follow-up procedures.
* Grade > or = 2 peripheral neuropathy.
* Any other malignancies within 5 years (except for treated carcinoma in situ of the cervix or basal cell skin cancer).
* Pregnant or lactating women ; patients with reproductive potential must use effective contraception.
* Inability to comply with follow-up procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 842 (Actual)
Dates: Start 2006-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival since randomization | time until progression

SECONDARY OUTCOMES:
Overall survival, | no time limit
toxicity (NCIC-CTC 3.0), | time until progression
quality of life (as assessed by LCSS). | until progression

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Pérol, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Maurice PEROL, Lyon, France

REFERENCES:
- [Result] Perol M, Chouaid C, Perol D, Barlesi F, Gervais R, Westeel V, Crequit J, Lena H, Vergnenegre A, Zalcman G, Monnet I, Le Caer H, Fournel P, Falchero L, Poudenx M, Vaylet F, Segura-Ferlay C, Devouassoux-Shisheboran M, Taron M, Milleron B. Randomized, phase III study of gemcitabine or erlotinib maintenance therapy versus observation, with predefined second-line treatment, after cisplatin-gemcitabine induction chemotherapy in advanced non-small-cell lung cancer. J Clin Oncol. 2012 Oct 1;30(28):3516-24. doi: 10.1200/JCO.2011.39.9782. Epub 2012 Sep 4. PMID 22949150